CLINICAL TRIAL: NCT05113628
Title: Methylene Blue Spray for Identification of Recurrent Laryngeal Nerve and Parathyroid Glands During Thyroidectomy: A Randomized Controlled Trial
Brief Title: Methylene Blue Spray for Identification of Recurrent Laryngeal Nerve and Parathyroid Gland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Methylene blue
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Methylene Blue; Recurrent Laryngeal Nerve Injuries; Parathyroid Gland
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anatomical identification (No Intervention): thyroidectomy was done with identification of both RLN and parathyroid gland done on anatomical basis
- methylene blue identification (Sham Comparator): thyroidectomy was done with identification of both RLN and parathyroid gland done using methylene blue spray (0.5 ml methylene blue 2% was diluted by 5ml normal saline) was sprayed over the lower thyroid pole and the perilobar area
  Interventions: Diagnostic Test: methylene blue identification

INTERVENTIONS:
Diagnostic Test: methylene blue identification — After ligation of the middle thyroid vein and the upper pole of the thyroid, the thyroid lobe was retracted medially and diluted methylene blue (0.5 ml methylene blue 2% was diluted by 5ml normal saline) was sprayed over the lower thyroid pole and the perilobar area. This area contains structures including recurrent laryngeal nerve, parathyroid glands, and inferior thyroid vessels which were observed After spraying.
  The vocal cord mobility was assessed intraoperatively by the anesthesiologist at time of extubation. The serum calcium was measured on the 2nd postoperative day. There was no routine use of postoperative calcium supplementation. Hypocalcemia was defined when the serum calcium level was less than 8 mg/dl.
  Arms: methylene blue identification

SUMMARY:
Thyroidectomy is the procedure by which surgeons treat various thyroid diseases and is considered the commonest endocrinal surgery. Yet, it carries a risk for intraoperative complications. The most distressing complications are recurrent laryngeal nerve and parathyroid injuries. Methylene blue spray is a technique than can be used for easy identification of both recurrent laryngeal nerve and parathyroid glands so we can avoid their injuries.

DETAILED DESCRIPTION:
Thyroid disorders constitute the second most common endocrine disease following diabetes mellitus. Thyroid surgery is one of the most frequently operated Head and Neck surgeries. Post-thyroidectomy complications are not uncommon. Parathyroids and Recurrent Laryngeal Nerve (RLN) are two of the complications of thyroidectomy that cause significant postoperative morbidity Due to the advances in thyroids surgeries, the occurrence of postoperative complications has been decreased, but when occurred, they cause lifelong handicap. The most important complications encountered are injury to the RLN and parathyroids. Meticulous dissection is a key factor in minimizing the occurrence of complications During thyroidectomy, careful dissection can protect the parathyroid glands and RLN. Various methods were used including capsular dissection, attention to protection of the arterial supply to parathyroids, avoiding unnecessary manipulation in the area of RLN Methylene blue spraying is a new technique that allows identification of both parathyroid glands and recurrent laryngeal nerves

ELIGIBILITY:
Inclusion Criteria:

* Age of 16 years and older.
* Both sexes.
* Patients who are candidate for thyroid surgery and euthyroid.

Exclusion Criteria:

* - Patients with hyper- or hypo-thyroid status.
* Patients who were unfit for surgery.
* Patients with unilateral or bilateral vocal cord palsy on preoperative indirect laryngoscopy
* Patients with thyroid malignancy by preoperative FNAC.
* Patients with hypersensitivity to methylene blue were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
detection of the recurrent larngeal nerve unstained | one minute after dye application
  the methylene blue dye stain the background and the RLN appears unstained
detection of the parathyroig glands | 3 minutes after dye application
  the methylene blue dye stain washed out and the parathyroid gland remained stained after 3 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university hospitals, Zagazig, Egypt